CLINICAL TRIAL: NCT03163368
Title: A Phase 1 Dose Escalation Trial of Neoadjuvant Radiosurgery for the Treatment of Metastatic Brain Tumors
Brief Title: Dose Escalation Trial of Neoadjuvant Radiosurgery for the Treatment of Metastatic Brain Tumors
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Stephen Shiao, Principal Investigator; Basic Science Director, Radiation Oncology, Cedars-Sinai Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT2016-18-Shiao-NeoAdSRS
Record Dates: First submitted 2017-05-19; First posted 2017-05-23 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-04

CONDITIONS: Brain Metastases
Keywords: metastatic tumor; brain lesion; stereotactic radiosurgery; neoadjuvant; maximum tolerated dose; dose escalation; neurosurgical resection
MeSH Terms: conditions — Brain Neoplasms; Neoplasm Metastasis | interventions — Craniotomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Neoadjuvant stereotactic radiosurgery (Experimental): Stereotactic radiosurgery will be performed prior to neurosurgical resection of the indexed brain metastasis. The dose of radiation to be administered to the indexed lesion will be established as a function of tumor size.
  Interventions: Radiation: Neoadjuvant stereotactic radiosurgery; Procedure: Neurosurgical resection

INTERVENTIONS:
Radiation: Neoadjuvant stereotactic radiosurgery — Dose escalation of neoadjuvant stereotactic radiosurgery
Procedure: Neurosurgical resection — Surgical resection of newly diagnosed brain metastases
  Other Names: craniotomy

SUMMARY:
The purpose of this study is to study if giving radiation to a brain tumor (a procedure called radiosurgery) before neurosurgery (surgery to remove the tumor) will help to keep brain tissue healthy, while possibly eliminating the need to return for radiation once a patient has healed from neurosurgery. This study will also seek the best radiation dose on a brain tumor based on how well the radiation therapy works and asses the side-effects.

DETAILED DESCRIPTION:
Radiosurgery is a non-surgical radiation therapy that can deliver targeted radiation to small brain tumors. Radiosurgery is considered to be part of standard of care. Typically for standard of care, radiosurgery is given after a patient has healed from neurosurgery, in an attempt to destroy any cancer cells that may be left after surgery. Patients who agree to participate in this research study will receive radiosurgery before their neurosurgery.

The timing of radiosurgery (pre-operatively) and the dosing to determine the safest dose is considered experimental.

By giving radiation the typical way, after surgery, a larger area of the brain must be covered, which means healthy brain tissue also receives radiation, whereas radiation before surgery will specifically target the tumor.

ELIGIBILITY:
Inclusion Criteria:

* Patients with prior histopathological diagnosis of cancer other than small cell lung cancer, lymphoma, and germ cell histologies.
* MR imaging of the brain with findings strongly suggestive of metastatic tumor(s) as assessed by the radiologist.
* MR evidence of at least one brain lesion ≤ 40 mm in maximal diameter that is deemed to be surgically resectable as evaluated by the neurosurgeon and appropriate for SRS. All other brain lesions must be appropriate for SRS alone and treated according to physician preference. Prior neurosurgery and/or prior SRS at a non-overlapping location are permitted at the discretion of the treating physician.
* Written informed consent obtained from subject, or a legally designated power of attorney and ability for subject to comply with the requirements of the study.
* Negative pregnancy test in women of childbearing potential (WOCBP) within 30 days of radiation. WOCBP is a female patient less than 50 years of age or who has menstruated within the last 12 months.
* Patients aged ≥ 18 years.
* Life expectancy ≥ 3 months
* Non-acute KPS ≥ 60%

Exclusion Criteria:

* Patients deemed medically unfit to undergo surgical resection of brain metastasis, such as those who are neurologically or hemodynamically unstable despite appropriate medical interventions.
* Patients who have had whole brain radiation within the previous three months.
* Patients with >4 brain metastases.
* Active or prior: documented inherited hypersensitivity syndromes, certain autoimmune diseases, and certain collagen vascular diseases. For example, any radiation hypersensitivity syndrome, including, but not limited to, ataxia-telangiectasia, Gorlin syndrome, multiple sclerosis, scleroderma, and systemic lupus erythematosus.
* Radiographic or cytologic evidence of leptomeningeal disease.
* Patients receiving methotrexate, adriamycin, epirubicine, or navelbin for one week prior to or concurrently with SRS. Note: All other systemic anti-cancer therapies will be reviewed on a case-by-case basis by study PI to determine if appropriate for study treatment and documented within the research record or EMR.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2017-05-09 (Actual); Primary Completion 2022-12-15 (Actual); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) | 1 month after neurosurgery
  To determine the maximum tolerated dose of radiosurgery given prior to neurosurgery in subjects with brain metastases of up to 4 cm.

SECONDARY OUTCOMES:
Adverse events | 1 month after neurosurgery
  To describe the adverse events associated with radiosurgery when administered prior to neurosurgical resection of brain metastases.
Describe preliminary rates of image-complete resection | 3 years
Describe preliminary rates of local tumor control | 3 years
Describe preliminary rates of intracranial control | 3 years
Describe preliminary rates of progression-free survival | 3 years
Describe preliminary rates of leptomeningeal spread | 3 years
Describe preliminary rates of rate of salvage treatment | 3 years
  Salvage treatment is any additional local treatment (surgery or radiation) in the setting of recurrent or progressive disease after the current treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Shiao, MD, PhD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No